CLINICAL TRIAL: NCT00556283
Title: Outcomes of Stapled Trans-Anal Rectal Resection (STARR) vs. Biofeedback in the Treatment of Outlet Obstruction Associated With Rectal Intussusception and Rectocele: A Multi-center Randomized Controlled Trial
Brief Title: RCT: STARR vs Biofeedback
Acronym: ODS II
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Ethicon Endo-Surgery (Europe) GmbH (Industry)
Collaborators: Aysgarth Statistics (Unknown); Physicians World GmbH (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ODS-HJH-4
Record Dates: First submitted 2007-11-08; First posted 2007-11-09 (Estimated); Last update posted 2013-12-18 (Estimated); Status verified 2013-12

CONDITIONS: Gastric Outlet Obstruction; Rectocele; Intussusception; Anismus
Keywords: outlet obstruction; rectocele
MeSH Terms: conditions — Gastric Outlet Obstruction; Rectocele; Intussusception | interventions — Biofeedback, Psychology

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): STARR
  Interventions: Device: STARR
- 2 (Active Comparator): Biofeedback
  Interventions: Behavioral: Biofeedback

INTERVENTIONS:
Device: STARR — Stapled Trans-Anal Rectal Resection for the treatment of ODS
  Arms: 1
Behavioral: Biofeedback — electromyographic-based treatment sessions
  Arms: 2

SUMMARY:
This study aimed to evaluate the safety and symptomatic outcomes achieved with Stapled Transanal Rectal Resection (STARR) compared to biofeedback training in patients with obstructed defecation syndrome (ODS).

ELIGIBILITY:
Inclusion Criteria:

1. Female patients >18 years old
2. Able to comprehend, follow, and provide written informed consent.
3. Minimum ODS Score of seven at screening.
4. Negative pregnancy test, by urine.
5. 'Obstructed' defecation requiring straining/digitation as presenting lead symptom.
6. Adequate external sphincter on rectal digital examination.
7. Evidence of anterior rectocele and/or rectal intussusception on dynamic defecography. (Note: dynamic defecography taken within 12 months will be acceptable)
8. Willingness to comply with study requirements including follow-up visits

Exclusion Criteria:

Evidence of external sphincter injury associated with incontinence.

1. Enterocele at rest- requiring surgery.
2. Faecal incontinence (soiling and faecal urgency is admissible).
3. Any anterior defect, colpocele or cystocele requiring a combined surgical approach.
4. Physical or psychological condition which would impair participation in the study.
5. Participation in any other device or drug study within 90 days prior to enrollment.
6. Planned participation in any other device study during the timeframe of this study.
7. General contraindication for surgery.
8. Previous transanal surgery for ODS.
9. Immunocompromised subjects

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 121 (Actual)
Dates: Start 2004-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
ODS total score | 12 months

SECONDARY OUTCOMES:
PAC-QoL score | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Lehur, MD, Principal Investigator — Institut des Maladies de l'Appareil Digestif (IMAD), University Hospital of Nantes, 1 place A Ricordeau, F-44093 Nantes Cedex 01; Goran Ribaric, MD, PhD, Study Director — Ethicon Endo-Surgery (Europe) GmbH
Locations (9):
- France (5):
  - Chirurgie Proctologique, Besançon
  - Clinique des Cèdres, Cornebarrieu
  - Groupe Hospitalier Diaconesses Croix Saint-Simon, Paris
  - Hopital Bagatelle, Talence
  - CHU Purpan, Toulouse
- Italy (3):
  - Ospedale S. Giuseppe, Milan
  - Ospedale "Franchini" di Montecchio Emilia, Montecchio Emilia
  - Ospedale Santa Maria degli Angeli, Pordenone
- Royal Liverpool University Hospital, Liverpool, United Kingdom